CLINICAL TRIAL: NCT06318754
Title: Large-bore Mechanical Thrombectomy for the Treatment of Symptomatic Portomesenteric Vein Thrombosis
Brief Title: Large-Bore Mechanic Thrombectomy for the Treatment of Symptomatic Portomesenteric Vein Thrombosis
Status: Withdrawn | Type: Observational
Why Stopped: PI is leaving UMB institution. IRB approval was never obtained and the study was never open.
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Inari Medical (Industry)
Responsible Party: Principal Investigator, Adam Fang, Assistant Professor of Diagnostic Radiology and Nuclear Medicine, University of Maryland, Baltimore
Other Study IDs: HP-00104241
Record Dates: First submitted 2024-02-23; First posted 2024-03-19 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-11

CONDITIONS: Thrombosis; Thrombectomy; Portal Vein
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Inari Triever Aspiration Catheter — Inari Triever Aspiration Catheter for portomesenteric venous thrombosis

SUMMARY:
A single site study evaluating the safety, feasibility, and effectiveness of percutaneous large-bore mechanical thrombectomy using the Inari Triever Aspiration Catheter for the treatment of portomesenteric vein thrombosis (PMVT).

DETAILED DESCRIPTION:
This is a single center, prospective, investigator-initiated observational study of adults undergoing mechanical thrombectomy as part of clinical care for portomesenteric vein thrombosis (PMVT).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years,
* PMVT diagnosed on cross-sectional imaging such as contrast-enhanced CT or MRI abdomen
* Symptomatic PMVT (persistent symptom, worsening abdominal pain after initiation of anticoagulation, development of peritonitis, complication of portal hypertension in cirrhosis (variceal bleeding or worsening ascites), and poor surgical candidates
* Speaks and understands English language

Exclusion Criteria:

* Age < 18 years
* no PMVT diagnosed on cross-sectional imaging such as contrast-enhanced CT or MRI abdomen
* Malignant PMVT
* chronic PMVT including presence of cavernoma and network of prominent collateral vessels in porta hepatis on cross-sectional imaging.
* asymptomatic PMVT
* life expectancy < 6 months
* Does not speak or understand English language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults undergoing a large-bore thrombectomy procedure for PMVT in the Division of Vascular and Interventional Radiology (VIR) at University of Maryland Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2025-03 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Technical Success | Time of intervention
  Uncomplicated transjugular access to the portal vein combined with uncomplicated implementation of the Inari Triever Aspiration Catheter for mechanical thrombectomy.
Clinical Success | 1 week, 1 month and 3 months post intervention
  Partial or complete resolution of patient's primary presenting symptoms, including ascites, gastrointestinal bleeding, and postprandial pain.
Primary Patency | 3 months post intervention
  Uninterrupted patency without any repeat intervention.
Intermediate functional success | Time of intervention
  Recanalization of the PMVT with re-established any level of hepatopetal flow in PMV system following Inari Flow Triever-assisted mechnical thrombectomy.

SECONDARY OUTCOMES:
Secondary Patency | 3 months post intervention
  Uninterrupted patency in patient who underwent re-intervention due to recurrent thrombosis.
Duration of hospitalization | 3 months post intervention
  Time from admission to hospital to the time of discharge from hospital.
Duration of ICU days | 3 months post intervention
  Time from transfer to ICU to discharge/transfer from ICU
Blood loss during intervention | At time of intervention
  Total amount of blood loss (mL) during the intervention
Transfusion | 3 months post intervention
  Total amount of PRBC given post-intervention and number of patient's requiring transfusion post-intervention.
Major and minor complications | 1 week, 1 month, and 3 months post intervention
  Society of Interventional Radiology major and minor complication will be used to categorize the complications.
30-day mortality | 30 days post intervention
  Death occurring within 30 days